CLINICAL TRIAL: NCT05064254
Title: Evaluating an Ultra-Brief Intervention for The Treatment Of COVID-19 Related Anxiety in Pregnant Women
Brief Title: Treatment of Anxiety in Pregnancy Study
Acronym: TAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other); Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TAPS
Record Dates: First submitted 2021-07-23; First posted 2021-10-01 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Anxiety; Pregnancy
Keywords: anxiety; pregnancy; pilot; brief psychotherapy; Mindfulness; virtual
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Single blind randomized controlled design. Pregnant women with anxiety symptoms will be randomly allocated 1:1 to either a control group (treatment as usual) or intervention group (treatment as usual plus MAPP intervention).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): All participants allocated to the control group will have access to standard care.
  Interventions: Other: Treatment as usual (TAU)
- Mindful Adaptive Practice in Pregnancy Therapy (Experimental): Participants allocated to the intervention group will have access to treatment as usual in addition to synchronous virtual MAPP.
  MAPP draws upon existing integrative principles of structured psychotherapies (mindfulness-based, cognitive, behavioural and relational psychotherapy)
  Interventions: Other: Treatment as usual (TAU); Other: Mindful Adaptive Practice in Pregnancy Therapy

INTERVENTIONS:
Other: Treatment as usual (TAU) — TAU may include self-help methods, physician visit, provision of resources etc.
Other: Mindful Adaptive Practice in Pregnancy Therapy — MAP teaches: a) recognition of personal maladaptive/ distressing patterns driving anxiety; b) how to relate differently; and c) cultivation of more adaptive ways of dealing with anxiety and learning how to effectively control it rapidly which allows re-engagement with life in more flexible ways.
  Other Names: MAPP
  Arms: Mindful Adaptive Practice in Pregnancy Therapy

SUMMARY:
Anxiety Disorders or Depressive Disorders with anxiety, affect about 3/5 pregnancies. It is known that if left untreated, these disorders are associated with poor delivery outcomes, ongoing mental illness, and negative effects on the child. The COVID-19 pandemic has created heightened anxiety in many people especially the most vulnerable. As a result, the investigators have seen that pregnant women report even higher rates of anxiety than in the past. Talk therapy is recommended but is underused in part because it takes a long time to learn and use. The COVID crisis has added another layer of complexity in that in-person treatment is not routinely available. The investigator team has adapted a talk therapy treatment, "Mindful adaptive practice in pregnancy (MAPP)" where women are taught skills to reduce anxiety. This treatment is done virtually over the internet in a synchronous group format. The overall objective of this study is to assess the feasibility, acceptability, and adherence to the clinical trial protocol evaluating MAPP on anxiety symptoms among pregnant women. This synchronous virtual treatment is novel and has the potential to change clinical practice as it will effectively reduce anxiety, takes a short time to learn and women will have access to it regardless of living in rural or remote areas. The results of this study will guide the development of a larger multi-site randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Antenatal mental illness is common. About 3/5 of women have antenatal anxiety or depression with anxiety which are both linked to adverse delivery outcomes and negative effects on child development. Often these conditions remain undetected/untreated, perpetuating the cycle of mental illness. A Canadian survey of pregnant women (~2000, April 2020) found >50% endorsed anxiety and > 2/3 elevated anxiety specific to pregnancy during the COVID-19 pandemic. This is on a background of elevated rates of antenatal mental illness. Psychotherapeutic interventions are preferred antenatally but barriers prevent their initiation and adherence (i.e., time duration). With the pandemic and the spike in anxiety, these vulnerable women are at risk to continue being ill and their child at risk for negative delivery/ longer-term outcomes. It is imperative these women receive rapid treatment to reduce acute anxiety to prevent mental health deterioration and the potential adverse effects. The pandemic has also forced clinicians to deliver healthcare in creative ways such as providing psychiatric care virtually despite their not knowing if the therapy can be effectively provided in this way and must be evaluated.

Mindful Adaptive Practice in Pregnancy (MAPP) is a novel ultra-brief psychotherapy developed by the investigator team to reduce anxiety. Prior work (nonclinical samples) suggested high recruitment and retention, significant distress reduction, and enhancement of wellbeing at rates comparable to gold standard therapies of longer duration. The work with clinical samples has shown it to have a large effect size. The investigators have adapted the technique to pregnant women to address the urgent clinical need for a brief, effective targeted intervention. As the investigators were challenged to offer health care services creatively, they adapted MAPP for virtual delivery, in a group format using the Ontario Telemedicine Network for example.

The overall objective of this study is to determine the feasibility, acceptability, and adherence to a clinical trial protocol evaluating the MAPP intervention on anxiety symptoms among pregnant women. The results of this pilot work will guide the development of a larger multi-site randomized controlled trial (RCT) to definitively evaluate the effectiveness of MAPP. As a secondary outcome, the investigators will assess the effect of MAPP in reducing anxious symptoms; this preliminary data on MAPP's effect will inform an effect size for the larger trial power analysis.

Pregnant participants from obstetrics, family practice, midwifery, and reproductive psychiatry clinics, as well as self-referral from social media, will be recruited. Sixty women will be randomized to the control group (standard care) or the intervention group (standard care plus MAPP). Outcomes will be captured electronically right after therapy ends, 3 months post-therapy, and 6 months post-therapy. Results of this work will be used for the larger trial which will have the potential to change clinical practice. Subsequent knowledge translation activities will foster knowledge uptake of the pilot results and once the final RCT is completed, the intervention will be widely disseminated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* >18 years of age
* At 12-30weeks gestation
* Score > 7 on the GAD-7
* Have internet access with camera, microphone, and ability to run the necessary software.
* Fluent in written and spoken English
* Willing to provide the name and contact details of their primary health care provider / other contact who would know person's whereabouts.

Exclusion Criteria:

* Current substance use
* Current psychotic/manic symptoms
* Active suicidal ideation
* Current use of psychotropic medication with dose change within 4 weeks of recruitment
* Currently receiving psychotherapy
* Unwilling to be randomized.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The number of participants screened positive for anxiety by the GAD-7 who are eligible for the study. | 11 months
  Among pregnant women who screen positive for anxiety, what is the rate of eligibility? The rate of eligibility will be determined as a raw percentage of the total number eligible over the total pool of participants entering the site.
The rate of recruitment as assessed by the number of participants recruited | 11 months
  Among eligible pregnant women who screen positive for anxiety, what is the rate of recruitment?
  The rate of recruitment will be determined as a raw percentage of the number recruited over the number eligible.
Reasons for non-participation as recorded by participants | 11 months
  Among pregnant women who screen positive for anxiety, what are the reasons for non-participation?
  Reasons for nonparticipation will also be calculated as a proportion.
Participant acceptability of treatment as measured by the Treatment Acceptability Scale | 6 weeks
  What are participants' level of perceived acceptability of the MAPP intervention?
  The Treatment Acceptability Scale (TAAS) will be used to assess participant acceptability of the intervention. It is a 10 item self report questionnaire where items were developed based on several factors including credibility, expectancy and perceived gaps specifically in the anxiety disorders literature. A 7-point Likert scale is used where higher scores indicate higher acceptability and anticipation to adhere to the intervention. The scale has good psychometric properties and is recommended for evaluating anxiety interventions.
Participant acceptability of treatment as measured by the Acceptability of Internet Delivery (AID)/ Experiences of Therapy Questionnaire | 6 weeks
  What are participants' level of perceived acceptability of the synchronous virtual group format?
  For the acceptability of internet delivery (AID), we will use questions that rate the importance of advantages and disadvantages of internet therapy in making a decision regarding using versus rejecting it.
Therapist acceptability of treatment as measured by the Acceptability of Intervention Measures | 6 weeks
  What are the therapists' perceptions of providing the MAPP intervention in a synchronous group format? For the acceptance of the virtual format, the therapists will complete the Acceptability of Intervention Measure (AIM) a four-item implementation measure that has been referred to as the "leading indicators" of successful implementation with shown psychometric strength and completion time being less than 1 minute.
Therapist acceptability of treatment as measured by questions on the Intervention Appropriateness Measure (IAM) | 6 weeks
  What are the therapists' perceptions of providing the MAPP intervention in a synchronous group format? For the acceptance of the virtual format, the therapists will complete the Intervention Appropriateness Measure (IAM), a four-item implementation measure that has been referred to as the "leading indicators" of successful implementation with shown psychometric strength and completion time being less than 1 minute.
Therapist acceptability of treatment as measured by the Feasibility of Intervention Measure (FIM) Questionnaire | 6 weeks
  What are the therapists' perceptions of providing the MAPP intervention in a synchronous group format? For the acceptance of the virtual format, the therapists will complete the Feasibility of Intervention Measure (FIM) a four-item implementation measure that has been referred to as the "leading indicators" of successful implementation with shown psychometric strength and completion time being less than 1 minute.
Participant Adherence to therapy as measured by proportion of participants who attend each session of therapy | 4 weeks
  What proportion of participants attend each session of therapy
  Proportion of participants completing each session over all participants for the session
Participant Adherence to therapy as measured by proportion of participants who attend all sessions of therapy | 4 weeks
  What proportion of participants all therapy session
  Proportion of participants completing all sessions over all participants
Participant Adherence to therapy as measured by the number completing follow-up questionnaires at 6, 12, and 24 weeks | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  What number complete all questionnaires at 6,12 and 24 weeks
  Proportion of participants over all at each time point
Participant Adherence to therapy as measured by recorded reasons for dropout | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  What are the reasons for drop out?
  Participants who drop out will be asked why and their answers will be recorded
Therapist Adherence to Therapy as assessed by therapist adherence checklists | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  What are the therapists' rate of adherence to the intervention? We will rate the therapists' adherence to the trial protocol by having independent assessors rate adherence by completing a checklist devised for the study intervention based on a previous successfully used framework. Comparisons will be made between therapists and their adherence rates

SECONDARY OUTCOMES:
Anxiety symptoms as measured by the GAD-7 | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  What is the effect of MAPP on anxiety symptoms compared to the control group at 6 weeks post randomization? The results from this question will be used to generate preliminary data on MAPP's effect on symptoms of anxiety compared to the control condition to inform an effect size for the larger trial power analysis. We will also assess at 12 and 24 weeks The GAD-7 is a 7-item anxiety scale with a min value of 0 and a maximum value of 21, with a higher score indicating higher levels of anxiety.

OTHER OUTCOMES:
Clinician rated anxiety as assessed by the Hamilton Anxiety Rating Scale (HAM-A) | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  Hamilton Anxiety Rating Scale (HAM-A) will be used as an objective measure of anxiety (to circumvent contamination of expectation) and completed prior to the other measures. The HAM-A is a 14-item, clinician-rated scale used to assess the severity of anxiety symptoms. Each item is rated on a 5-point likert scale where the total score ranges from 0 to 56. This scale shows good reliability, validity and sensitivity to change. Research staff blind to group will rate the items virtually.
Coronavirus anxiety as assessed by the COVID Anxiety Scale (CAS) | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  The COVID anxiety scale Assesses dysfunctional anxiety associated with the COVID-19 crisis. It has 5 items rated on a 0-4 Likert scale.
Participant Depression as assessed by the Edinburgh Postnatal Depression Scale The Edinburgh Postnatal Depression Scale (EPDS) | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  The Edinburgh Postnatal Depression Scale (EPDS) is an internationally recommended measure for depression symptoms in the perinatal period with well documented psychometric properties for pregnancy. Thirteen items are rated and a cutoff score > 12 will be used as recommended to identify depression.
Participant experiences of pregnancy as assessed by The Pregnancy Experiences Scale-Brief Version (PES-B) | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  The Pregnancy Experiences Scale-Brief Version (PES-B) will be used to measure overall pregnancy experience. It is made up of 10-items with positive and negative stressors specific to pregnancy rated from 0(not at all) to 3(great deal). Each item is rated on one dimension ("hassle or uplift"). We will calculate the intensity of hassles and uplifts (sum of scale scores (1-3)/hassles or uplift frequency. It has good reliability and validity for measuring positive and negative experiences.
Participant Healthcare Usage as assessed by the Edinburgh Health Care Utilization (HCU) | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  The Edinburgh Health Care Utilization (HCU) will be monitored to determine co-intervention or contamination. We will ask participants the number of visits they had with their psychiatrist, family physician for mental health reasons, and start of any treatments during the study period including medication. It has been used successfully in our previous studies with perinatal samples.
Participant Coping as assessed by the The Warwick Edinburgh Mental Well-being Scale (WMWS) | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  The Warwick Edinburgh Mental Well-being Scale (WMWS) will be used to measure coping skills. It consists of 14 positively worded items on scale of 0 to 5. Total scores range from 14 to 70 and it is psychometrically robust and used in pregnant women.
What is the effect of MAPP on pregnancy specific stressors | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  What is the effect of MAPP on pregnancy specific stressors
  The Pregnancy Related Anxiety Questionnaire R2 (PRAQ-R2) will capture pregnancy specific stressors. The 11 items of the PRAQ-R2 have strong evidence as pregnancy stressors.
What is the effect of MAPP on life stressors The Life Stress Inventory (LSI; Holmes & Rahe) general life stressors. The inventory is a well-known tool of 43 life events measuring stress load. | After therapy (4 weeks), 3 months post-therapy, and 6 months post-therapy
  What is the effect of MAPP on life stressors
Adverse effects | 6 weeks
  We will capture potential adverse effects by using a form made for the trial (Adverse effects form).
Demographics | Baseline
  Demographic information will be collected using a Socio-demographic questionnaire
Diagnoses | Baseline
  In order to better describe the sample, especially to be able to classify according to diagnosis, major psychiatric diagnoses will be captured with the Psychiatric Diagnostic Screening Questionnaire (PDSQ). It was developed to be a diagnostic aid in clinical practice and with current psychiatric nomenclature. It is self-report and assesses the most common major psychiatric diagnoses seen in outpatient mental health settings. It has good reliability and validity. While half of participants will randomly receive the PDSQ, the other half will be randomized to receive the Mini International Neuropsychiatric Interview (MINI) anxiety and depression modules. The purpose of using both questionnaires is to validate the PDSQ as an equivalent measurement to the MINI diagnostic inventory in our patient population and will use only the PDSQ for our future large
Therapists' activities log-intervention activities | 4 weeks
  Therapists' activities (session completed / date, telephone discussions if any, missed sessions etc.) will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Grigoriadis, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Center; Steven Selchen, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Center
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No